CLINICAL TRIAL: NCT02573116
Title: Impact of Treatment of Periodontis on Endothelial Function in Patients With Obstructive Sleep Apnea
Acronym: EndothSAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/44
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Disease in Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; endothelial dysfunction; periodontitis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obstructive sleep apnea with chronic parodontis (Experimental): patients with severe obstructive sleep apnea (OSA) and chronic parodontis treated for OSA by continuous positive airway pressure (CPAP) and intensive periodontal treatment
  Interventions: Procedure: scaling and root planing
- Obstructive sleep apnea without chronic parodontis (No Intervention): patients with severe OSA treated by CPAP

INTERVENTIONS:
Procedure: scaling and root planing — full-mouth intensive removal of subgingival dental plaque biofilms with the use of scaling and root planing after the administration of local anesthesia
  Arms: Obstructive sleep apnea with chronic parodontis

SUMMARY:
Evaluation of the add-on effect on endothelial dysfunction of treatment of periodontitis in patients with chronic periodontitis and severe obstructive sleep apnea treated by CPAP. Patients with and without chronic periodontitis will be treated by CPAP for 20 weeks. At V2 (10 weeks), endothelial dysfunction will be assessed by the Reactive Hyperemia- Peripheral Artery Tone index. The endothelial dysfunction of the patients will be also assessed at V3 (20 weeks) after periodontitis treatment for the group of patients with chronic periodontitis.

DETAILED DESCRIPTION:
At V2, patients with periodontitis will have full-mouth intensive removal of denatl plaque biofilms with the use of scaling and root planing. The add-on effect of the periodontitis treatment on endothelial dysfunction will be assessed ten weeks later (V3) in comparison with V2 by taking into account with the effect of 10 weeks of CPAP in the control group with severe OSA but not periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* severe OSA defined by an apnea hypopnea index > or = 30 per hour
* with or without chronic parodontitis

Exclusion Criteria:

* non equilibrated diabetes
* obesity (BMI > or = 40)
* active smoker (> 1 pack per day (20 cigarettes))
* pregnancy
* antibiotics within the preceding three months
* prophylactic antibiotherapy required for the parodontitis treatment
* acute parodontitis or all parontal pathology requiring immediate therapy
* less than 10 teeth

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 20 weeks
  measure of Reactive Hyperemia- Peripheral Artery Tone index with Endopat

SECONDARY OUTCOMES:
Endothelial function | 10 weeks
  measure of Reactive Hyperemia- Peripheral Artery Tone index with Endopat
blood biomarkers | 0, 10 and 20 weeks
  hsCRP, leptin, adiponectin, E-selectin and orosomucoid
Epworth Sleepiness Scale | 0, 10 and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Henno, MD, Principal Investigator — AP-HP, Hôpital Européen Georges Pompidou
Locations (1):
- Hôpital Foch, Suresnes, France